CLINICAL TRIAL: NCT06397534
Title: The Effect of the Flipped Learning Model on the Knowledge and Self-Efficacy Level of Nursing Students Regarding Stoma Care: A Randomized Controlled Study
Brief Title: Flipped Learning Model on the Stoma Care
Acronym: Stomacare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Ankara Yildirim Beyazit University, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FlippedLearningModel
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Stoma Colostomy; Nursing Caries; Nursing Student
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped Learning (Experimental): In the experimental group, students will be administered the "Introduction Characteristics Form," "Stoma Care Knowledge Assessment Form (pre-test)," and the "General Self-Efficacy Scale (pre-test)." Subsequently, digital materials (such as stoma care presentation materials and stoma care demonstration videos) will be prepared by the researchers. The video content will be uploaded to the 'Edpuzzle' program, which is accessible via internet connection or downloadable to devices. The video content in the 'Edpuzzle' program will consist of stoma care procedural steps. Following this, students will apply the "stoma care" skill in the skills laboratory under the supervision of instructors. To reinforce the implementation in the experimental group, online activities such as word clouds and quizzes will be sent. After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.
  Interventions: Other: Education
- Control (No Intervention): All students in the control group will be administered the 'Introductory Characteristics Form,' the 'Stoma Care Knowledge Assessment Form (pre-test),' and the 'General Self-Efficacy Scale (pre-test).' Subsequently, stoma care will be provided to the control group solely through traditional teaching methods. No additional resources will be provided. The stoma care topic will be taught to the control group for 2 hours theoretically and for 4 hours practically. Teaching in the control group will be conducted through PowerPoint presentations, question-and-answer sessions, demonstrations, and discussions. After the lesson, students will practice 'stoma care' in the skills laboratory under the supervision of instructors. After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.

INTERVENTIONS:
Other: Education — In the experimental group, students will be administered the "Introduction Characteristics Form," "Stoma Care Knowledge Assessment Form (pre-test)," and the "General Self-Efficacy Scale (pre-test)." Subsequently, digital materials (such as stoma care presentation materials and stoma care demonstration videos) will be prepared by the researchers. The video content will be uploaded to the 'Edpuzzle' program, which is accessible via internet connection or downloadable to devices. The video content in the 'Edpuzzle' program will consist of stoma care procedural steps. Following this, students will apply the "stoma care" skill in the skills laboratory under the supervision of instructors. To reinforce the implementation in the experimental group, online activities such as word clouds and quizzes will be sent. After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.
  Arms: Flipped Learning

SUMMARY:
This study is planned as a randomized controlled trial to determine the effect of education provided through the flipped learning model on students' levels of knowledge and self-efficacy regarding stoma care. The research will be conducted on 100 first-year nursing students between 05.2024-06.2024. Randomization will be ensured for students who meet the inclusion criteria, and they will be divided into two random groups: the experimental group (n=50) and the control group (n=50). All participating students will be administered the "Introductory Characteristics Form," "Stoma Care Knowledge Assessment Form (pre-test)," and "General Self-Efficacy Scale (pre-test)." For students in the experimental group, digital materials required for preparedness for the course based on the flipped learning model (such as course presentation materials and demonstration videos) will be prepared by the researchers. After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.

All students in the control group will be administered the 'Introductory Characteristics Form,' the 'Stoma Care Knowledge Assessment Form (pre-test),' and the 'General Self-Efficacy Scale (pre-test).' Subsequently, stoma care will be provided to the control group solely through traditional teaching methods. No additional resources will be provided.

After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.

DETAILED DESCRIPTION:
The Effect of the Flipped Learning Model on the Knowledge and Self-Efficacy Level of Nursing Students Regarding Stoma Care: A Randomized Controlled Study Introduction In nursing education, where theoretical and applied education is provided as a whole, students are expected to acquire cognitive, affective, and psychomotor skills. Within this education, students are expected to become proficient in some fundamental clinical skills. One of these skills that students are expected to acquire is stoma care. It is important for students to learn stoma care correctly before going into clinical practice, and they are expected to perform these skills flawlessly. Proper implementation of the steps of stoma care is crucial. When stoma care is not performed correctly, serious complications such as bleeding, infection, peristomal skin problems, stoma ischemia, and necrosis may occur in patients (Aşti & Karadağ, 2021; Berman et al., 2008; Lynn et al., 2011). These types of complications lead to prolonged hospital stays and increased costs for patients. Minimizing the occurrence of such complications in patients is essential for improving their adaptation to stoma, reducing their distress, enhancing their quality of life, and ensuring the comfort of future clinical nurses, who will provide effective care. Therefore, it is seen that stoma care holds an important place in the nursing process, and it needs to be learned competently in educational life.

It is crucial to teach stoma care correctly and to impart this skill in nursing education. Therefore, different teaching methods can be used to teach stoma care in nursing education. One of these teaching methods is the flipped learning model. The flipped learning model is a pedagogical approach that involves providing students with pre-class information about the topic to be covered and facilitating learning through interactive activities with students during class (Herreid & Schiller, 2013). This approach was proposed as the Flipped Classroom concept by Bergmann and Sams (2012). This method, which provides students with rich learning opportunities and ensures that they come to class prepared, engages students actively in the learning process during class. In a flipped classroom, instructors support students in learning the information they have learned, discuss unclear topics, and engage students in active learning activities (Bergmann & Sams, 2012; Critz & Knight, 2013). This model is an innovative and effective practice that provides students with both individually personalized and group learning environments (Aksoy, 2020).

There is no research found in the literature evaluating the effect of the flipped learning approach on nursing students' knowledge and self-efficacy in stoma care. In this context, it can be said that evaluating the subject of stoma with the flipped learning approach will reflect on the learning and teaching experiences of both students and educators. This research is planned to determine the effect of education provided with the flipped learning model on stoma care knowledge and self-efficacy levels.

Materials and Methods Study Design This study is planned as a randomized controlled experimental study. Hypotheses: H1: The flipped learning model increases students' knowledge of stoma care. H2: The flipped learning model enhances students' self-efficacy regarding stoma care.

Study Location and Characteristics The research will be conducted at the Faculty of Health Sciences, Department of Nursing, Ankara Yıldırım Beyazıt University.

Population and Sample of the Study This study will be conducted during the spring semester of the 2023-2024 academic year at the Faculty of Health Sciences, Department of Nursing, Ankara Yıldırım Beyazıt University. The Principles of Nursing Course is taught during the spring semester (8 hours theory and 16 hours practice). The theoretical content of the courses is delivered through lectures, question-answer sessions, and discussions by the instructors. In addition to theoretical knowledge, practical skills are developed through demonstrations and laboratory work in areas where psychomotor skills need to be improved. Clinical applications begin after theoretical education and laboratory work. Stoma care is taught for two hours theoretically and four hours in the laboratory.

The population of the study will consist of 190 first-year students enrolled in the Faculty of Health Sciences, Department of Nursing, Ankara Yıldırım Beyazıt University during the 2023-2024 academic year.

Students who are enrolled for the first time in the Principles of Nursing course, volunteer to participate in the research, and have access to a smartphone/computer and continuous internet usage will be included in the study. Students who have previously studied in a health-related field and have previously taken the Principles of Nursing course will be excluded from the study.

Sample size calculation was conducted with G-Power 3.1.9.7 statistical software. A total of 100 students, with 50 in the experimental group and 50 in the control group, are required based on a power analysis using the mean knowledge scores from a similar study (Cohen, 1992), considering a 5% error margin, an effect size of 0.57, and a power level of 80%.

Data Collection Tools The data of the study will be collected using the "Demographic Characteristics Form," "Stoma Care Knowledge Evaluation Form" (pre-test-post-test), and "General Self-Efficacy Scale." Demographic Characteristics Form (Form 1): This form, prepared by the researchers, consists of 4 questions regarding students' demographic characteristics (age, gender, frequency of computer use, frequency of smartphone use).

Stoma Care Knowledge Evaluation Form (pre-test-post-test) (Form 2): This form includes 20 statements related to stoma care, such as what a stoma is, the characteristics of a stoma, emptying a stoma bag, changing a stoma bag, and skin care around the stoma. The statements were developed based on the literature (ASCN Stoma Care Clinical Guidelines 2016, Tuzer, Elbas, 2016). Each statement is evaluated on a 100-point scale, with options for "Correct," "Incorrect," and "I don't know." Correct responses are scored as 1, incorrect responses as 0, and the total score is calculated out of 100. 12 statements are correct and 8 statements are incorrect.

General Self-Efficacy Scale (Form 3): The scale, developed by Sherer et al. (1982) and validated and reliability-tested in Turkish by Yıldırım and İlhan (2010), consists of three sub-dimensions and 17 items. The scale's sub-dimensions include "Starting" (items 2, 4, 5, 6, 7, 10, 11, 12, and 17; min-max: 9-45), "Persistence" (items 3, 13, 14, 15, and 16; min-max: 5-25), and "Effort Sustainment-Insistence" (items 1, 8, and 9; min-max: 3-15). The scale is a 5-point Likert-type scale, with response options ranging from "5: describes me very well" to "1: does not describe me at all" for each item. The scale includes 11 reverse-scored items (items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, and 17). The maximum score that can be obtained from the scale is 85 and the minimum score is 17. An increase in score indicates an increase in self-efficacy belief.

Implementation of the Study Randomization will be ensured for the students participating in the research, dividing them into two random groups: the experimental group and the control group. All students who meet the inclusion criteria will undergo the administration of the "Demographic Characteristics Form," "Stoma Care Knowledge Evaluation Form (pre-test)," and "General Self-Efficacy Scale (pre-test)." Experimental Group: For students in the experimental group, digital materials required for preparedness for the course based on the flipped learning model (such as course presentation materials and demonstration videos) will be prepared by the researchers. The video content in the 'Edpuzzle' program will consist of stoma care procedural steps. The video content in the 'Edpuzzle' program will consist of stoma care procedural steps. Following this, students will apply the "stoma care" skill in the skills laboratory under the supervision of instructors. To reinforce the implementation in the experimental group, online activities such as word clouds and quizzes will be sent. After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.

Control Group: All students in the control group will be administered the 'Introductory Characteristics Form,' the 'Stoma Care Knowledge Assessment Form (pre-test),' and the 'General Self-Efficacy Scale (pre-test).' Subsequently, stoma care will be provided to the control group solely through traditional teaching methods. No additional resources will be provided. The stoma care topic will be taught to the control group for 2 hours theoretically and for 4 hours practically. Teaching in the control group will be conducted through PowerPoint presentations, question-and-answer sessions, demonstrations, and discussions. After the lesson, students will practice 'stoma care' in the skills laboratory under the supervision of instructors. After the implementation and 4 weeks later, the 'Stoma Care Knowledge Assessment Form (post-test)' and the 'General Self-Efficacy Scale (post-test)' will be administered online.

After the laboratory application of the control and experimental groups, the "Stoma Care Knowledge Evaluation Form (post-test)" and "General Self-Efficacy Scale (post-test)" will be administered.

Data Analysis: The collected data will be analyzed using SPSS 15 software. The normal distribution of the data will be evaluated using the Kolmogorov-Smirnov test. Independent samples t-test will be used to determine differences between groups, repeated measures analysis of variance (ANOVA) will be used for dependent triple groups (pre-test-post-test-follow-up), and paired t-test will be used to determine the means that differ in the three groups.

Permission obtained from the Ankara Yıldırım Beyazıt University Ethics Committee and the Faculty of Health Sciences, Department of Nursing for the implementation of the research. Students will be informed about the research and their consent will be obtained. Permission has been obtained for the use of the General Self-Efficacy Scale.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing students,
* Volunteer to participate in the research,
* Have smartphones/computers
* Have continuous Internet Access

Exclusion Criteria:

* Have previously studied in a health-related field
* Have previously taken the fundamentals of nursing course

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-17 (Estimated); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Stoma Care Knowledge Evaluation Form | just before education, just after education, just 1 month after education
  This form includes 20 statements related to stoma care, such as what a stoma is, the characteristics of a stoma, emptying a stoma bag, changing a stoma bag, and skin care around the stoma. The statements were developed based on the literature (ASCN Stoma Care Clinical Guidelines 2016, Tuzer, Elbas, 2016). Each statement is evaluated on a 100-point scale, with options for "Correct," "Incorrect," and "I don't know." Correct responses are scored as 1, incorrect responses as 0, and the total score is calculated out of 100. 12 statements are correct and 8 statements are incorrect.
General Self-Efficacy Scale | just before education, just after education, just 1 month after education
  The scale, developed by Sherer et al. (1982) and validated and reliability-tested in Turkish by Yıldırım and İlhan (2010), consists of three sub-dimensions and 17 items. The scale's sub-dimensions include "Starting" (items 2, 4, 5, 6, 7, 10, 11, 12, and 17; min-max: 9-45), "Persistence" (items 3, 13, 14, 15, and 16; min-max: 5-25), and "Effort Sustainment-Insistence" (items 1, 8, and 9; min-max: 3-15). The scale is a 5-point Likert-type scale, with response options ranging from "5: describes me very well" to "1: does not describe me at all" for each item. The scale includes 11 reverse-scored items (items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, and 17). The maximum score that can be obtained from the scale is 85 and the minimum score is 17. An increase in score indicates an increase in self-efficacy belief.

IPD SHARING:
Plan to Share IPD: No